CLINICAL TRIAL: NCT07214064
Title: Safety and Feasibility of a Venetoclax- Augmented Treosulfan-Based Reduced Intensity Conditioning Before Allogeneic Stem Cell Transplantation in AML, MDS/AML and Higher Risk MDS
Brief Title: Venetoclax- Augmented Treosulfan-Based Reduced Intensity Conditioning Before Allogeneic Stem Cell Transplantation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VeStAL; 2025-521372-62-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: AML (Acute Myeloid Leukemia); MDS/AML; MDS (Myelodysplastic Syndrome)
Keywords: Allogeneic Stem Cell Transplantation; Venetoclax; Venetoclax- Augmented Treosulfan-Based Reduced Intensity Conditioning; RIC
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced Intensity Conditioning before Allogeneic Stem Cell Transplantation (Experimental): Patients with AML, MDS/AML or HR-MDS, who have either responded to remission inducing therapy or are intended for upfront transplantion receive conditioning chemotherapy as follows:
  IMPs:
  * Venetoclax 400 mg abs. day -8 to day -2
  * Fludarabine 30 mg/m2 BSA day -6 to day -2
  * Treosulfan 10 g/m2 BSA day -4 to day -2
  Interventions: Drug: RIC regimen

INTERVENTIONS:
Drug: RIC regimen — Venetoclax (Venclyxto®): 400 mg abs./d day -8 to -2, Fludarabine 30 mg/m2 BSA day -6 to day -2, Treosulfan 10 g/m2 BSA day -4 to day -2

SUMMARY:
Safety and Feasibility of a Venetoclax- Augmented Treosulfan-Based Reduced Intensity Conditioning Before Allogeneic Stem Cell Transplantation in AML, MDS/AML and Higher Risk MDS

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years at the time of signing the Informed Consent
2. Patient is fluent in German
3. Signed written Informed Consent with the cognitive ability to understand all consequences of trial participation and to comply with all trial related procedures
4. Diagnosis of AML,MDS/AML (according to ICC 20226) or HRMDS (IPSS-R7 >3.5 or IPSS-M8 >0; according to ICC 20226 and IWG 20232)
5. Myeloid neoplasm (AML, MDS/AML or HR-MDS according to ICC 20226) under control* at time of screening, defined as one of the following:

   5.1. AML (ICC 20226):

   • Scheduled for alloHCT after prior Remission

   Induction ± Consolidation:
   * Achievement of at least MLFS** (according to ELN 20221 criteria) after up to two cycles of intensive, anthracycline-based induction chemotherapy OR
   * Achievement of at least MLFS** (according to ELN 20221 criteria) after intensive, anthracycline-based induction chemotherapy folllowed by up to three cycles of cytostatic consolidation therapy OR
   * Achievement of at least MLFS** (according to ELN 20221) after less intensive, HMA-based treatment (up to six cycles) OR
   * Achievement of at least MLFS** (according to ELN 20221) after a combination of intensive and less intensive treatments (up to six cycles in total) 5.2. MDS/AML (ICC 20226):• Scheduled for alloHCT after prior Remission

   Induction ± Consolidation:
   * Achievement of at least MLFS** (according to ELN 20221 criteria) after up to two cycles of intensive, anthracycline-based induction chemotherapy OR
   * Achievement of at least MLFS** (according to ELN 20221 criteria), after intensive, anthracycline-based induction chemotherapy folllowed by up to three cycles of cytostatic consolidation therapy OR
   * Achievement of at least MLFS** (according to ELN 20221 criteria) after less intensive, HMA-based treatment (up to six cycles and including HMA monotherapy) OR
   * Achievement of at least MLFS (according to ELN 20221 criteria) after a combination of intensive and less intensive treatments (up to six cycles in total)• Scheduled for upfront alloHCT:
   * ≤19% bone marrow blastsAND• ≤19% peripheral blood blastsAND• ≤15.000/µl peripheral blood Leukocytes 5.3. HR- MDS (ICC 20226, IWG 20232)
   * Scheduled for alloHCT after prior therapy:
   * up to six cycles of a less intensive HMAbased treatment or HMA monotherapy AND
   * ≤9% bone marrow blastsAND• ≤9% peripheral blood blasts• Scheduled for upfront alloHCT:
   * ≤9% bone marrow blasts AND
   * ≤9% peripheral blood blasts *The disease is considered clinically controlled, when it is either aggressive but has proven responsive to cytostatic chemotherapy (e.g. AML with achievement of at least MLFS) or slowly progressive ( e.g. suitable for upfront alloHCT in cases of MDS/AML) or is both slowly progressive and responsive to therapy

     * a bone marrow assessment is mandatory during screening phase. Patients canonly be enrolled after the according inclusion criteria have been confirmed bybone marrow biopsy. The time window for bone marrow biopsy is day -21 to -14.
6. Eligiblity for alloHCT according to a board of experienced haematologists
7. Karnofsky Performance Index ≥60%
8. Planned alloHCT with Peripheral Blood Stem Cells (PBSC)
9. Infusion of allogeneic stem cells schedulded between day 14 and day 28 after Screening
10. Availability of a suitable donor, defind as one of the following:

    10.1. HLA-identical sibling (MSD)OR 10.2. HLA-compatible (9/10 antigens matched for HLA-A, -B, -C, -DRB1, and -DQB1) unrelated donor (MUD) with completed confirmatory typing.

    OR 10.3. Two unrelated donors with >90% probability of a 9/10 match for HLA- A, -B, -C, -DRB1, and -DRQB1, according to OptiMatch list (MUD)
11. Documented diffusion lung capacity for carbon monoxide (DLCO) >40% (adjusted for hemoglobin, if available) and FEV1/FVC >50%
12. Left ventricular ejection fraction (LVEF) ≥40%
13. GFR (CKD-EPI) ≥ 30 ml/min/1,73 m2
14. Bilirubin ≤3x ULN and AST ≤5x ULN
15. Thoracic imaging (either X-ray or computed tomography (CT)) without evidence of active infection or second malignancy
16. Subject (male or female) is willing to use highly effective methods during treatment and for 6 months (male or female) after the end of treatment (adequate: combined hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner1, sexual abstinence2). Female participants using homonal contraceptives should use a barrier method as well.1 Vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the FCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success2 In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
17. Absence of pregnancy confirmed by a highly sensitive pregnancy test not older than 3 days at time of screening (only FCBP).
18. Subject agrees not to share medication.

Exclusion Criteria:

1. APL (AML with t(15;17))
2. MDS/MPN (ICC 20226)
3. Karnofsky Performance Index <60%
4. Patient scheduled for haploidentical allogeneic hematopoetic stem cell transplantation or bone marrow stem cell transplantation
5. Presence of extramedullary myelosarcoma
6. Disease Relapse after prior CRc
7. History of allogeneic hematopoietic stem cell transplantation
8. Significant active cardiac disease within 6 months prior to the start of study treatment, including:

   * New York Heart Association (NYHA) class III or IV congestive heart failure
   * Myocardial infarction
   * Unstable angina
   * Cerebral apoplexy
   * Severe cardiac arrhythmias
   * Left ventricular ejection fraction (LVEF) <40% by TTE
9. Documented diffusion lung capacity for carbon monoxide (DLCO) ≤40% (adjusted for hemoglobin, if available) and FEV1/FVC ≤50%
10. GFR (CKD-EPI) <30 ml/min/1,73 m2
11. Bilirubin >3x ULN or AST >5x ULN
12. Clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia.
13. Active viral infection, including hepatitis B, hepatitis C or Human Immunodeficiency Virus (HIV) infection, that is uncontrolled prior to first dose of study treatment and may interfere with the study objectives or which could expose the patient to undue risk through the participation in the clinical trial. An infection controlled with an approved antiviral treatment is allowed.
14. Presence of Proven, Probable or Possible Invasive Fungal Disease (IFD) as defined by EORTC/MSG 20209 Definitions (please consult Appendix)
15. Serologies suggestive of recent (<6 months) infection or reactivation with/of Toxoplasma gondii (based on IgG, IgM and Avidity) or of infection with Treponema pallidum (based on TPPA).
16. Any clinically uncontrolled infection (bacterial or unknown pathogen), defined as persisting or recurring fever or rising levels of CRP (≥10 mg/dl) despite intravenous antibacterial or antifungal therapy (initiated or escalated at least 72h hours ago)
17. Immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding and/or disseminated intravascular coagulation.
18. Conditions that limit the ingestion or gastrointestinal absorption of orally administered drugs.
19. Patients with a currently active second malignancy. Patients are not considered to have a currently active malignancy, if they have completed therapy and are considered by their physician to be at <30% risk of relapse within one year. However, patients with the following history/concurrent conditions are allowed:

    * Basal or squamous cell carcinoma of the skin;
    * Carcinoma in situ of the cervix;
    * Carcinoma in situ of the breast;
    * Incidental histologic finding of prostate cancer.
20. Receipt of live, attenuated vaccine within 30 days prior to the study inclusion (NOTE: patients, if enrolled, should not receive live vaccine during the study and until 6 months after the therapy)
21. Severe neurological or psychiatric disorder interfering with ability to give an informed consent.
22. Women during pregnancy and lactation.
23. History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
24. Participation in other trials interfering with the endpoint of this study. Prior trial participation is permitted, provided that treatment with the investigational medicinal product has been completed at least 4 days prior to screening for this trial (at least 10 days before planned study treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | at day 28 after alloHCT
  Primary objective of this trial is to evaluate the feasibility and safety of the augmentation of a treosulfanbased RIC regimen for alloHCT in AML, MDS/AML and HR-MDS patients with the Bcl-2-inhibitor Venetoclax. As outlined above, the aim is to increase antileukemic acitiviy without increasing morbidity and mortality in a vulnerable patient collective. This is operationalized by the following primary endpoint:
  1) Overall survival (OS) at day 28 after alloHCT Most adverse events (AEs) due to the IMPs are expected to occur before day 0. Protacted or lateonset toxicities with potentially lethal consequences cannot be ruled out. Therefore, we regard it most suitable to evaluate overall survival at day 28 after alloHCT.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Faul, Dr., Principal Investigator — Sponsor's Delegate
Locations (1):
- University Hospital , Department of Internal Medicine II, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No